Assessing Inflammatory and Behavioral Pathways Linking PTSD to Increased Asthma Morbidity in WTC Workers

PI: JuanWisnivesky MD NCT04552301

Document Date: 9/21/2021

**Icahn School of Medicine at Mount Sinai** 

## 

Form Version Date: 09/21/20

### STUDY INFORMATION:

Study Title: Assessing Inflammatory and Behavioral Pathways Linking PTSD to Increased Asthma

Morbidity in WTC Workers: Phase II

Principal Investigator (Head Researcher): Juan P. Wisnivesky, MD, DrPH

Physical Address: 17 E. 102nd St., D6-119, New York, NY 10029

Mailing Address: One Gustave L Levy Place Box 1087, NY, NY

Phone: 212-824-7567

### **SUMMARY OF THIS RESEARCH STUDY:**

In medicine there are many unanswered questions. A research study is when scientists try to answer a question about something that we don't know enough about. Participation in a research study may or may not directly help you or others. Participation is entirely voluntary. It is completely up to you whether or not you take part. You can also change your mind at any time and it will not affect your ability to get medical care within the Mount Sinai Health System.

The purpose of this study is to develop and test a program for asthma and Post-Traumatic Stress Disorder (PTSD) by adapting Cognitive Processing Therapy (CPT) with asthma education for individuals who were affected by the World Trade Center (WTC) disaster. CPT is a PTSD treatment that focuses on how the traumatic event is understood and coped with by a person who is trying to regain a sense of mastery and control in his or her life.

If you choose to participate, you will be asked to attend 10 1-hour weekly in-person, teleconference, or phone sessions, and 3 research interviews (1 interview before starting the pilot and 2 follow-up interviews after completing the pilot at 1 week and 3 months). You will be asked to participate in discussions with a Study Interventionist about your experiences during and after the World Trade Center disaster and your asthma management. If you are unable to attend any of the sessions, you will be given the opportunity to complete up to 1 make up sessions individually with the Study Interventionist. There are no costs associated with participation in this pilot and you will be compensated for your time and effort.

The main risks to you if you choose to participate are minimal.

You may not benefit from participation in this study. You may also benefit from participation in this research by developing improved health and self-management behaviors.

If you are interested in learning more about this study, please continue to read below.

FOR IRB USE ONLY ev 1.16.19

Effective Date: 9/21/2021

End Date:9/20/2022

Icahn School of Medicine at Mount Sinai


### PARTICIPATION IN THIS RESEARCH STUDY:

This research study will be fully explained to you by a member of the study team. Feel free to ask all the questions you want before you make a decision about whether or not to participate. Any new information that develops during this research study that might make you change your mind about participating will be given to you promptly.

You may qualify to take part in this research study because you are at least 18 years of age, may have PTSD based on the Structured Clinical Interview for DSM-IV (SCID), speak English, have been diagnosed with asthma by a healthcare provider, take an asthma controller medication, and have participated in the observational phase of the Assessing Inflammatory and Behavioral Pathways Linking PTSD to Increased Asthma Morbidity in WTC Workers study.

Funds for conducting this research are provided by Centers for Disease Control and Prevention (CDC).

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

### LENGTH OF TIME AND NUMBER OF PEOPLE EXPECTED TO PARTICIPATE:

Your participation in this research study is expected to last 24 weeks.

The number of people expected to take part in this research study at the Icahn School of Medicine at Mount Sinai is 40.

### **DESCRIPTION OF WHAT'S INVOLVED:**

If you agree to participate in this research study, the following information describes what may be involved.

- You will be asked to attend 10 1-hour weekly in-person, teleconference, or phone sessions with a Study Interventionist.
- You will be asked to participate in discussions related to your experiences before, during and after the World Trade Center disaster that may have contributed to PTSD symptoms.
- You will be asked to participate in discussions related to your asthma management behaviors.
- You will be asked to have your asthma medication with you in each session.
- You will be asked to complete an initial interview (baseline) before you meet with the study interventionist.
- You will be asked to complete a follow-up interview at 1 week and 3 months after you complete the
  pilot sessions during which you will be asked to answer questions about your asthma, disease
  beliefs and self-management behaviors.

FOR IRB USE ONLY

ev 1.16.19

Effective Date: 9/21/2021 End Date: 9/20/2022 Icahn School of Medicine at Mount Sinai

## ****


- You will be either be in the Cognitive Processing Therapy (CPT) and tailored asthma education group or to the Supportive Psychotherapy and general asthma education group.
- The CPT group focuses on how the traumatic event is understood and coped with by a person who is trying to regain a sense of mastery and control in his or her life. The asthma components that will be integrated into the intervention include psychoeducation about asthma, barriers to asthma selfcare, asthma medication education, inhaler technique, and asthma self-management behaviors.
- The Supportive Psychotherapy group will be given emotional support and general education on managing asthma.
- The sessions may be conducted in person, over the phone, or through teleconference.
- Your sessions may be recorded for quality improvement. These recordings will not be identified to
- The study treatment you get will be chosen by chance, like flipping a coin. You have an equal chance of being in either group, but will know which group you have been assigned to.

# **USE OF YOUR DATA:**

In the future, your identifiable information may be removed from the private information that if collected as part of this research. After this removal, the information could be used for future research studies or shared with other research teams for future research studies. You will not be informed of the details of specific research that is done with your medical information. That means that a research project might be done that you would not consent to if provided with the details of that research project.

The researchers would like to ask your permission to keep the data collected from you during this study to use them in future research studies. Please tell us how we may use this material in future research studies.

| (1) Will you all studies? | ow the researd | hers to store your information to use in future research |
|---|---|---|
| Yesnext question. | | If no, please stop here. If yes, please continue to the |

(2) The researchers can keep your information stored in one of two different ways: one way will store your information and/or specimens in a way that it is linked to your identity (through the use of a code that can indicate the information came from you personally) and the other way will store your information and/or specimens anonymously (no one will know who the information is from). It will not be stored both ways, so you must choose one of these two options. Please note that if you choose to have your information and/or specimens stored anonymously, you will not be able to change your mind to ask for your information and/or specimens to be destroyed at a future date. How would you like your information and/or specimens stored? Please initial **ONE** choice:



End Date:9/20/2022

FOR IRB USE ONLY

Effective Date: 9/21/2021

**Icahn School of Medicine at Mount Sinai** 

# 

|---|
| I would like my information stored with a link to my identity I would like my information stored anonymously |
| (3) Do you give the researchers permission to <b>contact you</b> in the future to collect additional information about you, discuss how your information might be used, or to discuss possible participation in another research project? Please initial your choice: |
| YesNo |
| (4) Do you give the researchers permission to keep the information indefinitely and use them for future studies that are <b>directly related</b> to the purpose of the current study? Please initial your choice: |
| YesNo |
| (5) Do you give the researchers permission to keep the information indefinitely and use them for future studies that are <b>not related</b> to the purpose of the current study (for example, a different area of research)? Please initial your choice: |
| YesNo |
| <b>(5.1)</b> From time to time researchers outside of medicine and related sciences would like to use this information. This might be in the field of anthropology, human origins, mapping human migration patterns etc. Do you give permission to use your information outside the fields of medicine and biological sciences? Please initial your choice: |
| YesNo |
| (a) If the future research in a different area can be done without having to know that the information came from you personally, that will be done. (b) If the future research in a different area requires that it is known specifically who the information and/or specimens came from, then one of the following will be done: (i) If you allowed the researchers to contact you in the future, they may be able to contact you to explain why your identifiable information is needed and what will be done with it. Your permission will be asked to use your information in that research project. (ii) If you do not give permission to be contacted in the future, or if it is found that contacting you is not practical, for example, because you have moved, your identifiable data may still be used. The Institutional Review Board (IRB) will be asked for permission to use the information and/or specimens linked to your identity. The IRB can give permission for researchers to use and share identifiable health information without contacting you, but only if it determines that sharing the information will not be more than a minimal risk to you or your privacy. The Institutional Review Board (IRB) is a committee of doctors and scientists and nonscientists, including people not associated with this hospital or medical school, whose job it is to protect people who participate in research. |

FOR IRB USE ONLY

IRB Approved ev 1.16.19

Effective Date: 9/21/2021

End Date:9/20/2022

Icahn School of Medicine at Mount Sinai

## 


| (6) Do you give permission to have portions of the information given to other researchers, i | ncluding |
|---|---|
| those at Mount Sinai, other academic institutions and for profit companies, for use in research | ch within |
| the limits you have chosen above? Please initial your choice: | |

| Yes No |
|--------|
|--------|

### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study you will be responsible for the following things:

- Attending sessions
- Completing brief homework assignment provided by the Study Interventionist, if applicable
- Having your asthma medications during the sessions
- Completing the follow-up interview at the end of the pilot

### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

If you agree to take part in this research study, we will pay you up to \$290 for your time and effort. You will receive \$20 for each completed Pilot session (up to \$200 total) and \$30 for completing the each interview. All payments will be made in the form of cash or money order depending on whether the visit is completed in-person, through teleconference, or over the phone.

| Pilot Study | Payment |
|---------------------|--------------------|
| Pilot Baseline | \$30 |
| Per Session | \$20 (total \$200) |
| 1 Week Follow-Up | \$30 |
| 3 Month Follow-Up | \$30 |
| Total (Pilot Study) | \$290 |

Tax law may require the Mount Sinai Finance Department to report the amount of payment you receive from Mount Sinai to the Internal Revenue Service (IRS) or other agencies, as applicable. Generally, this reporting would take place if you receive payments that equal \$600 or more from Mount Sinai in a calendar year. You would be responsible for the payment of any tax that may be due.

FOR IRB USE ONLY



Effective Date: 9/21/2021 End Date:9/20/2022 Icahn School of Medicine at Mount Sinai


| <b>Form</b> | Version | Date: | 09/21/20 |
|-------------|---------|-------|----------|
|-------------|---------|-------|----------|

#### **POSSIBLE BENEFITS:**

It is important to know that you may not get any benefit from taking part in this research. Others may not benefit either. However, possible benefits may be improved health knowledge and health behaviors.

### **REASONABLY FORESEEABLE RISKS AND DISCOMFORTS:**

Your participation will involve minimal risks or discomforts.

- Psychological risks (for example, embarrassment, fear or guilt). You are not required to answer any questions that make you feel uncomfortable. The Study Interventionist implementing the intervention will be trained in a variety of therapeutic approaches. If a participant remains upset or wishes to speak to another individual, a clinical psychologist, social worker or qualified medical professional will be sought in those cases.
- Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

### OTHER POSSIBLE OPTIONS TO CONSIDER:

You may decide not to take part in this research study without any penalty. The choice is totally up to you.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY:

If you believe that you have suffered an injury related to this research as a participant in this study, you should contact the Principal Investigator.

### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this research study at any time without any penalty. This will not affect your ability to receive medical care at any of the Mount Sinai Health System hospitals or to receive any benefits to which you are otherwise entitled.

If you decide to stop being in the research study, please contact the Principal Investigator or the research staff.

If you decide you don't want your data to be used for research anymore, you can contact the researcher and ask to have your data removed from future use. If any data have already been shared without your identity, it won't be possible to retrieve them because no one will know who you are. Data that have already been used will not be affected by your decision. Any data that are still linked to your

FOR IRB USE ONLY

ev 1.16.19

Effective Date: 9/21/2021 End Date: 9/20/2022 Icahn School of Medicine at Mount Sinai

## 


identity by a code the researcher has will be withdrawn so that no future sharing of your samples and/or data will take place.

<u>Withdrawal without your consent</u>: The study doctor, the sponsor or the institution may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the study team have not been followed, the investigator believes it is in your best interest, or for any other reason. If data have been stored as part of the research study, they too can be destroyed without your consent.

#### **CONTACT INFORMATION:**

If you have any questions, concerns, or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Principal Investigator at 212-824-7567.

This research has been reviewed and approved by an Institutional Review Board. You may reach a representative of the Program for Protection of Human Subjects at the Icahn School of Medicine at Mount Sinai at telephone number (212) 824-8200 during standard work hours for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research subject.
- You want to get information or provide input about this research.

### **DISCLOSURE OF FINANCIAL INTERESTS:**

Sometimes, physicians/researchers receive payments for consulting or similar work performed for industry. Effective September 2014 Mount Sinai reviews only payments to an individual totaling more than \$5,000 a year per entity when determining potential conflicts of interest. If you have questions regarding industry relationships, we encourage you to talk your physician/researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

### **MAINTAINING CONFIDENTIALITY - HIPAA AUTHORIZATION:**

As you take part in this research project it will be necessary for the research team and others to use and share some of your private protected health information. Consistent with the federal Health Insurance Portability and Accountability Act (HIPAA), we are asking your permission to receive, use and share that information.

FOR IRB USE ONLY

IRB Approved

Effective Date: 9/21/2021 End Date: 9/20/2022 Icahn School of Medicine at Mount Sinai

**Icahn School of Medicine at Mount Sinai** 

### 


What protected health information is collected and used in this study, and might also be shared with others?

As part of this research project, the research team at the hospital(s) involved in the research will collect your name, address, phone number, date of birth, age and medical record number.

The researchers will also get information from your medical record from the Mount Sinai Health System.

During the study the researchers will gather information by:

- Taking a medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.

### Why is your protected health information being used?

Your personal contact information is important to be able to contact you during the study. Your health information and the results of any tests and procedures being collected as part of this research study will be used for the purpose of this study as explained earlier in this consent form. The results of this study could be published or presented at scientific meetings, lectures, or other events, but would not include any information that would let others know who you are, unless you give separate permission to do so.

The Principal Investigator may also use and share the results of these tests and procedures to treat you in collaboration with others in the Mount Sinai Health System.

The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example, the School's Program for the Protection of Human Subjects is responsible for overseeing research on human subjects, and may need to see your information. If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes. If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

### Who, outside Mount Sinai, might receive your protected health information?

As part of the study, the Principal Investigator, study team and others in the Mount Sinai workforce may disclose your protected health information, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Principal Investigator.)

- Other collaborating research center(s) and their associated research/clinical staff who are working with the investigators on this project: University of Colorado, Denver and the Hospital for Sick Children and other sites available on request.
- The sponsoring government agency and/or their representative who need to confirm the accuracy of the results submitted to the government or the use of government funds: NHLBI

FOR IRB USE ONLY

ev 1.16.19

Effective Date: 9/21/2021 End Date:9/20/2022 Icahn School of Medicine at Mount Sinai

**Icahn School of Medicine at Mount Sinai** 

## 


- A Data Safety Monitoring Board or other committee that will monitor the study on an ongoing basis for safety.
- The United States Department of Health and Human Services and the Office of Human Research Protection.

In almost all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier. Some records and information disclosed may be identified with a unique code number. The Principal Investigator will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the Institutional Review Board allows it after determining that there would be minimal risk to your privacy. The Certificate of Confidentiality obtained from the Department of Health and Human Services will not be used to prevent disclosure to local authorities of child abuse and neglect, or harm to self or others. It is possible that a sponsor or their representatives, a data coordinating office, or a contract research organization, will come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, the Office of Human Subjects Protection (OHRP) of the Department of Health and Human Services as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. They are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. We may publish the results of this research. However, we will keep your name and other identifying information confidential.

For how long will Mount Sinai be able to use or disclose your protected health information?: Your authorization for use of your protected health information for this specific study does not expire.

### Will you be able to access your records?

During your participation in this study, you will not be able to access your medical records. This will be done to prevent the knowledge of study results from affecting the reliability of the study. Your information will be available should an emergency arise that would require your treating physician to know this information to best treat you. You will have access to your medical record and any study information that is part of that record when the study is over or earlier, if possible. The investigator is not required to release to you research information that is not part of your medical record.

Do you need to give us permission to obtain, use or share your health information?

NO! If you decide not to let us obtain, use or share your health information you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment or enrollment in any health plans or affect your eligibility for benefits.

### Can you change your mind?

You may withdraw your permission for the use and disclosure of any of your protected information for research, but you must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, the Principal Investigator for the research study may still use your protected information that was already collected if that information is necessary to complete the

FOR IRB USE ONLY



Effective Date: 9/21/2021 End Date: 9/20/2022 Icahn School of Medicine at Mount Sinai

**Icahn School of Medicine at Mount Sinai** 

## 


study. Your health information may still be used or shared after you withdraw your authorization if you should have an adverse event (a bad effect) from being in the study. If you withdraw your permission to use your protected health information for research that means you will also be withdrawn from the research study, but standard medical care and any other benefits to which you are entitled will not be affected. You can also tell us you want to withdraw from the research study at any time without canceling the Authorization to use your data.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, even if your information will no longer be protected by federal regulations, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If as part of this research project your medical records are being reviewed, or a medical history is being taken, it is possible that HIV-related information may be revealed to the researchers. If that is the case, the following information concerns you. If this research does not involve any review of medical records or questions about your medical history or conditions, then the following section may be ignored.

### **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 306-5070. These agencies are responsible for protecting your rights.

### Certificate of Confidentiality:

To further protect your privacy, the researchers have obtained a Certificate of Confidentiality from the Department of Health and Human Services. This is intended to ensure that your identity as a participant in this research study will not have to be disclosed as a result from a subpoena, for the purpose of identifying you in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings other than to the FDA or OHRP as identified above.

The research staff will not share any of your research information or biospecimens with anyone who is not a member of the research team, including any family members or friends, other than to those identified above. However, you should know that if we learn that you or someone else is threatened with serious harm, such as a child or an elderly person being abused, the investigators may notify the appropriate authorities if necessary to protect you or others. A Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research. This means that you and your family must also actively protect your own privacy. If an insurer or employer learns about your research participation, and you agree that they can have your research information, then the researchers may not use the Certificate of Confidentiality to keep this information from them.

FOR IRB USE ONLY

ev 1.16.19

Effective Date: 9/21/2021 End Date: 9/20/2022 Icahn School of Medicine at Mount Sinai

# 


| Signature of subject | Printed Name of Subject | Date | Time |
|---|---|---|---|
| PERSON EXPLAINING STUDY | AND OBTAINING CONSENT: | | |
| | Printed Name of consent delegate | | — — Time |
| Signature of consent delegate | 3 | | |
| WITNESS SECTION:<br>When a witness is required to ob-<br>example, when subject is illiterate | serve the consent process, it should be<br>e, visually impaired, or this document ac | | |
| example, when subject is illiterate<br>consent).<br>My signature below documents th | serve the consent process, it should be | ccompanies<br>nent and ar | a short form or a short form |

FOR IRB USE ONLY

ev 1.16.19

Effective Date: 9/21/2021 End Date:9/20/2022 Icahn School of Medicine at Mount Sinai